CLINICAL TRIAL: NCT05246384
Title: A Phase I/Ib, Open-label Study to Evaluate the Safety, Pharmacokinetics and Clinical Activity of RP7214, a Dihydro-orotate Dehydrogenase (DHODH) Inhibitor, Administered Orally in Combination With Azacitidine in Patients With Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Acute Myeloid Leukemia
Brief Title: Study to Evaluate the Safety, Pharmacokinetics and Clinical Activity of RP7214 in Combination With Azacitidine in Patients With Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia and Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in development plan
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP7214-2102
Record Dates: First submitted 2022-01-29; First posted 2022-02-18 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia
Keywords: RP7214; Dihydro-orotate Dehydrogenase (DHODH)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — RP7214

STUDY DESIGN:
Intervention Model Description: open-label, non-randomized, two-part Phase I/Ib study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I (dose escalation) RP7214 + Azacitidine (Experimental): Participants will receive RP7214 orally in combination with Azacitidine in a 28-day cycle. The dose levels will be escalated until MTD/a recommended Phase 2 dose (RP2D) has been identified.
  Interventions: Drug: RP7214
- Part II (dose expansion) RP7214 + Azacitidine (Experimental): Participants will receive RP7214 orally at the MTD/RP2D in combination with Azacitidine in a 28-day cycle.
  Interventions: Drug: RP7214

INTERVENTIONS:
Drug: RP7214 — RP7214 will be administered daily twice a day orally; Azacitidine will be administered from Days 1 to 7 of each 28-day cycle

SUMMARY:
This is a multi-center, open-label, non-randomized, two-part Phase I/Ib study of RP7214 in combination with azacitidine in patients with AML, MDS and CMML. Part I is a 3+3 dose-escalation study to identify the MTD/RP2D of RP7214 and azacitidine combination in patients with AML, MDS, and CMML. Part II is a dose-expansion study to evaluate the clinical activity and safety of RP7214 and azacitidine combination in AML.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must sign informed consent.
2. Patient should be ≥ 18 years of age.
3. Patients who are candidates for treatment with azacitidine and present with one of the following:

   a. Part I: Dose Escalation study i. Patient with histologically or cytologically confirmed relapsed/refractory AML as per World Health Organization (WHO) classification, 2016 'OR' ii. Newly diagnosed AML patients who are ineligible for intensive induction chemotherapy due to co-morbidity or other factors 'OR' iii. Intermediate-2 or high-risk MDS according to the International Prognostic Scoring System (IPSS) 'OR' iv. Chronic Myelomonocytic Leukemia (CMML) b. Part II: Dose Expansion study i. Newly diagnosed AML patients who are ineligible for intensive induction chemotherapy due to co-morbidity or other factors.
4. Patient should have an Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2.
5. Patients must be amenable to serial bone marrow biopsies/aspirates and peripheral blood sampling as required by the protocol.

Exclusion Criteria:

1. Any cancer-directed therapy taken (e.g., chemotherapy, immunotherapy, biologic therapy or an investigational drug) within 14 days or 5 half-lives, whichever is shorter, prior to C1D1. For radiation therapy, at least 60 days should elapse from prior Total Body Irradiation (TBI) and at least 14 days from local palliative radiation therapy.
2. Patients with rapidly increasing peripheral blast counts (WBC count > 25,000/μL) while on hydroxyurea prior to C1D1.
3. Patients with Acute Promyelocytic Leukemia (French American-British Class M3 AML).
4. Patients on immunosuppressive therapy post autologous or allogeneic stem cell transplantation (ASCT or Allo-SCT) at the time of screening, or with clinically significant Graft-Versus-Host Disease (GVHD) in the opinion of the Investigator or has not recovered from transplant-associated toxicities prior to C1D1.
5. Patient who discontinued prior therapy with DHODH inhibitors or azacitidine due to drug-related toxicity.
6. Evidence of uncontrolled/progressing infection.
7. Patients with immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or Disseminated Intravascular Coagulation (DIC).
8. Presence of isolated extramedullary relapse.
9. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of RP7214 in combination with azacitidine | 28 days
  The maximum tolerated dose will be defined as the highest dose tested in which a DLT is experienced by 0 out of 3 or 1 out of 6 patients among the dose levels.

SECONDARY OUTCOMES:
Tmax | 35 days
  Pharmacokinetics: Time to Reach Maximum Concentration (Tmax) of RP7214
Objective Response Rate (ORR) | 2 years
  Defined as the percentage of patients who achieve Complete Remission (CR), Complete Remission with incomplete bone marrow recovery (CRi) and Partial Remission (PR)
Clinical Benefit Rate (CBR) | 2 years
  Defined as the percentage of patients achieving a CR, CRi, PR and Stable Disease (SD) lasting for at least 8 weeks.
Duration of Remission | 2 years
  Defined as the number of days from the date of first remission (CR, CRi, or PR) to the recurrence or Progressive Disease (PD)
Percentage of patients requiring blood and/or platelet transfusions | 2 years
  Defined as number of patients requiring blood and/or platelet transfusions
Cmax | 35 days
  Pharmacokinetics: Maximum Concentration (Cmax) of RP7214
AUC | 35 days
  Pharmacokinetics: Area Under the Concentration Curve (AUC) of RP7214

IPD SHARING:
Plan to Share IPD: No